CLINICAL TRIAL: NCT05708521
Title: Optimization of Post-Operative Pain Following Orthognathic Surgery With Personalized Opioid Prescription and Tapering Protocols
Brief Title: Personalization of Opioid Prescription Following Orthognathic Surgery
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Amr Alsabbagh, Resident in Oral and Maxillofacial Surgery, Masters Graduate Student, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 52007
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Pain, Postoperative; Orthognathic Surgery; Opioid Use; Patient Satisfaction; Opioid Use Disorder
Keywords: Personalized Opioid Prescription; Opioid Tapering Protocol; Orthognathic Surgery; Post-Operative Pain; Patient Satisfaction
MeSH Terms: conditions — Pain, Postoperative; Patient Satisfaction; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to one of 2 parallel study arms and followed longitudinally. Their allocation to the study arms will be performed by using a random number generator, whereby if the number 0 arises, they are allocated to the control group, and if the number 1 arises, they are assigned to the experimental group.
Who Masked: Participant
Masking Description: Participants will be masked to which group they are assigned to avoid the placebo effect.
  Given the nature of the study in which opioid prescription quantities are controlled and questionnaires provide a detailed schedule of opioid dosage and frequency, providers and investigators cannot be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standardized Prescription Group (SOP) (Active Comparator): All participants assigned to the SOP group will be treated as per the current status quo, in which they are given the standardized analgesic prescriptions following discharge from the hospital consisting of:
  1. Acetaminophen 975 mg orally every 6 hours for 7 days
  2. Ibuprofen 600 mg orally every 6 hours for 7 days
  3. Hydromorphone 2-4 mg orally every 6 hours as needed, with a total dispense amount of 40mg.
  The participants are not given instructions on how to taper their hydromorphone medication, which is the current status quo in our department.
  Interventions: Drug: Standardized dose and frequency of hydromorphone with no tapering post-orthognathic surgery
- Personalized Prescription Group (POP) (Experimental): All participants assigned to the POP group will receive pre-operative education on the medications that they will be given while they are inpatients and upon discharge, along with a pain medication card to aid their understanding. Medications upon discharge will be:
  1. Acetaminophen 975mg orally every 6 hours for 1 week
  2. Ibuprofen 600 mg orally every 6 hours for 1 week
  3. Hydromorphone - Prescribed with a personalized schedule and tapering protocol based on the participant's last 24-hour in-patient use of opioids.
  Participants in this arm will also receive tapering instructions as well as an education card to assist them with their tapering protocol upon discharge.
  Interventions: Drug: Personalization of dose and frequency and instituting a tapering protocol of hydromorphone post-orthognathic surgery

INTERVENTIONS:
Drug: Personalization of dose and frequency and instituting a tapering protocol of hydromorphone post-orthognathic surgery — POP participants will be given a personalized opioid prescription with a tapering protocol based on their last inpatient 24-hour usage of opioids, obtained from the nursing medication administration record. Should a participant stay in the hospital for less than 24 hours (e.g. patient had an early discharge at 18 hours), the 24-hour in-patient opioid usage would be extrapolated from their total amount and frequency of opioid use. The participant will be provided with an instruction card with suggestions on how much opioid to take at various time points following discharge to safely taper their medication.
  Arms: Personalized Prescription Group (POP)
Drug: Standardized dose and frequency of hydromorphone with no tapering post-orthognathic surgery — SOP participants will be given a standardized dose of hydromorphone (2-4mg orally every 6 hours), and a total amount of 40mg. No further information is provided to them with regards to their pain medication and to tapering.
  Arms: Standardized Prescription Group (SOP)

SUMMARY:
This study aims to investigate pain management and satisfaction following orthognathic surgery, which is a type of surgery that corrects jaw and facial bone issues. This type of surgery can result in significant post-operative pain for participants, and the goal of this study is to find a way to manage this pain in a more effective and safe manner.

The study will focus on the use of opioid pain medication and will compare two groups: one group will receive a standardized prescription plan. In contrast, the other group will receive a personalized prescription with a plan to taper the opioid medication. In the end, any unused opioid will be compared at the end of the 7-day post-discharge period between the two groups. This is important because excessive opioid prescription can either be diverted to the community or can be misused leading to opioid use disorders.

Data will be collected from pre-surgery appointments, during the surgery and hospital stay, and follow-up appointments. The data collected will include participants' demographics, medical history, type of surgery, and information about the pain medication used.

The study hypothesizes that the personalized prescription plan will result in less unused medication and higher satisfaction with pain management compared to the standardized prescription plan. The study will also stratify the participants into single-jaw surgery and double-jaw surgery groups to evaluate if any differences in the outcomes are observed. This study will help to provide guidance for future pain management practices for participants undergoing orthognathic surgery. Furthermore, this study will also benefit society by providing insights into addressing the opioid crisis that is currently affecting many communities across North America.

DETAILED DESCRIPTION:
This study aims to investigate the use of post-operative pain management following orthognathic surgery, with a focus on the use of opioid medication. Orthognathic surgery is a foundational surgery for the correction of dentofacial deformities, which requires osteotomies, rearrangement, and fixation of the facial bones into a new position. Participants are often placed into maxillomandibular fixation postoperatively, limiting the range of motion of the mandible. The surgical trauma provoked by the osteotomies, stripping of facial muscles, and swelling of the associated soft tissue envelope can result in significant post-operative pain in participants. This pain is one of the primary reasons participants are admitted following surgery for up to several days. Further complicating pain management for these participants is the maxillomandibular fixation, which reduces the ability of participants to verbally communicate with their nursing staff about their levels of pain.

Multimodal analgesia using a combination of acetaminophen, non-steroidal anti-inflammatory drugs (NSAIDs), and opioid medications are the mainstay therapies for acute post-surgical pain. However, long-term opioid use can lead to opioid tolerance, due to various mechanisms, including receptor desensitization and downregulation. This can lead to persistent postoperative opioid use and opioid use disorder.

In Canada, the opioid crisis is on the rise in all provinces, driven by both illegal and prescription opioids. Most opioid-related deaths occurred in males between the ages of 30 to 39, with an overall increase in the use rate amongst younger age groups. Canada has the second highest rate of opioid prescription in the world, after the United States of America. The legitimate use of opioid analgesics in adolescents - who otherwise disapprove of illegal drug use - is independently associated with a 33% increased risk of opioid misuse in later life. Furthermore, persistent opioid use may be the most common complication after elective surgery. Currently, in our department, much like many other oral and maxillofacial surgical centers, there is a "standardized" prescription of opioids, such as hydromorphone, for all participants being discharged from the hospital. However, it is clear from the literature and anecdotal evidence that most participants do not require as much opioids as we currently prescribe.

In the last few years, there have been recent initiatives to personalize post-operative pain management in orthopedic joint replacement as well as spine surgeries. In these studies, the primary consideration for opioid dosing and frequency following discharge relies on the participants' opioid requirements while in the hospital. A tapering protocol and cessation timeline following discharge is tailored for each participant based on their in-patient opioid requirements to promote opioid prescription stewardship further. These studies demonstrated a reduction in post-operative opioid consumption, with no changes in perceived pain and participants' satisfaction.

This study aims to assess the postoperative analgesic efficacy, opioid requirement, and total analgesic requirements for participants undergoing orthognathic surgery with a personalized discharge opioid prescription and tapering protocol. The study will compare two groups of participants: one group will receive the standardized prescription plan of hydromorphone, while the other group will receive a personalized prescription plan. The control will receive a standardized discharge prescription of 2-4 milligrams of liquid hydromorphone taken orally every 4 hours as needed for pain, with a total prescription of 40 milligrams of hydromorphone. The experimental group will receive a personalized hydromorphone prescription and tapering protocol for the study group. This prescription will be inferred from the participant's last 24-hour in-patient requirement of opioids before being discharged. The personalized schedule is based on a modification of a prescription schedule for spine and orthopedic joint procedures derived by Dr. Edward Mariano's group at Stanford University's Department of Anesthesiology, Perioperative and Pain Medicine.

Data will be obtained from the pre-admission appointment, and in-patient records including the nursing medication administration record (MAR), intra-operative anaesthesia records, participants' questionnaires, and the first follow-up appointment at 2 weeks. Data collected will include the participant's age, weight, body mass index, sex, pertinent medical and psychiatric history, pre-surgical anxiety, type of orthognathic surgery, length of surgery, length of stay in the hospital, amount and frequency of analgesics taken by the participants while in-hospital, analgesic dosages prescribed to the participants on discharge, amount and frequency of analgesics taken by the participants for each day following discharge, remaining prescribed opioids at the 2-week follow-up appointment, and the participant's self-reported satisfaction and pain on the Defense and Veterans Pain Rating Scale (DVPRS) questionnaire. All patient questionnaires will be recorded via REDCap, a secure online data management software.

Subjects will be stratified into single jaw surgery (i.e. LeFort only, BSSO only, +/- FG), or double jaw (i.e. LeFort and BSSO +/- FG). A Mann-Whitney U Test will be utilized for statistical analysis, with significance assumed at p < 0.05. This study is important as it will help to provide guidance for future pain management practices for participants undergoing orthognathic surgery and also help promote opioid stewardship.

ELIGIBILITY:
Inclusion criteria

1. Patients undergoing orthognathic surgery for the correction of dentofacial deformities. Included in the study will be patients who receive single-jaw surgery (i.e. BSSO [Bilateral Sagittal Split Osteotomy, a surgery of the lower jaw] only, or Lefort [osteotomy of the upper jaw] only), or those in the double-jaw surgery category (BSSO and Lefort).
2. Patients undergoing a functional genioplasty who have an additional osteotomy included in their surgical plan (i.e. BSSO and/or Lefort).
3. Patients undergoing cleft orthognathic surgery.

Exclusion criteria

1. Patients who are under the age of 18 at the time of surgery
2. Patients who are contraindicated to undergo elective surgery, including pregnant patients.
3. Patients with a history of opioid use disorder.
4. Patients on chronic opioids within the past month.
5. Patients who have a contraindication for multimodal analgesia (e.g. renal injury precluding the prescription of NSAIDs).
6. Patients with allergies to opioids, acetaminophen, and/or NSAIDs.
7. Patients receiving a surgically-assisted rapid palatal expansion (SARPE) surgery due to the different post-operative nature of the surgery.
8. Patients who have previously undergone prior orthognathic (i.e. repeat surgery), non-cleft craniofacial surgery, or have previously experienced maxillofacial trauma due to the potential alterations in neural pain pathways.
9. Patients undergoing an isolated functional genioplasty.
10. Patients who are unable to consent to surgery and/or the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Fraction (%) of remaining unused opioid | Assessed at 7-days post-discharge, which is the point at which participant would have completed their post-operative recovery period and are expected to have ceased using their prescribed opioid medication.
  The participant will self-report how much liquid hydromorphone (1mg/mL) remains in millilitres after they have stopped consuming it for management of their acute post-surgical pain, expected to be at 7-days post-op. The participant will also bring their remaining opioid to their first follow-up appointment to confirm this measurement.
  The remaining opioid is compared to their prescribed opioid to determine the relative amount of unused opioid measured as a percentage.
Absolute amount (milligrams) of remaining unused opioid | Assessed at 7-days post-discharge, which is the point at which participant would have completed their post-operative recovery period and are expected to have ceased using their prescribed opioid medication.
  The participant will self-report how much liquid hydromorphone (1mg/mL) remains in millilitres after they have stopped consuming it for management of their acute post-surgical pain, expected to be at 7-days post-op. The participant will also bring their remaining opioid to their first follow-up appointment to confirm this measurement.
  The remaining opioid is compared to their prescribed opioid to determine the absolute amount of unused opioid measured in milligrams.

SECONDARY OUTCOMES:
Overall satisfaction with post-surgical pain management at home | Assessed at the 7-day post-discharge period, which is the point at which participants would have completed their post-operative recovery period and are expected to have used most of their prescribed opioid medication.
  The participant's overall satisfaction with their post-surgical pain management at home as measured on the supplemental questions in the Defense and Veterans Pain Rating Scale questionnaire.
  The scale measures the participants satisfaction by asking them to indicate a score from 0 to 10 for 4 items on how the pain: interferes with activity, interferes with sleep, affects overall mood, and contributes to overall stress.
  A score of 0 indicates that the pain does not contribute or interfere with the aforementioned items (i.e. patient is very satisfied), while a score of 10 indicates significant contribution or interference (i.e. patient is very dissatisfied).
Mean duration of usage of opioids | Assessed at the 7-day post-discharge period, which is the point at which participants would have completed their post-operative recovery period and are expected to have used most of their prescribed opioid medication
  The secondary outcome measure is the mean duration of usage of opioids measured in number of days used post-operatively.
Total daily use of opioid by the participant | Assessed at the 7-day post-discharge period, which is the point at which participants would have completed their post-operative recovery period and are expected to have used most of their prescribed opioid medication
  Measured as total morphine milli-equivalents (MME) per day from the questionnaire filled out by the participant. Information is cross-referenced with the total remaining opioid brought back at the follow-up visit.
Average daily pain scores following discharge | Assessed at the 7-day post-discharge period, which is the point at which participants would have completed their post-operative recovery period and are expected to have used most of their prescribed opioid medication
  The participant indicates their level of pain each time they take an analgesic medication following discharge from hospital. This is based on the Defense and Veterans Pain Rating Scale, where a score of 0 indicates no pain, while a score of 10 indicates that the pain is severe.
  The average of the scores for each day is obtained and reported as the average daily pain score.

CONTACTS AND LOCATIONS:
Overall Officials: Amr Alsabbagh, DDS, Principal Investigator — Dalhousie University; Jean-Charles Doucet, DMD, MD, MSc, Study Chair — Dalhousie University
Locations (1):
- Dalhousie University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make the individual participant data (IPD) collected in this study available to other researchers. This decision was made to protect the privacy of the participants involved in the study and to ensure that their personal information is not shared without their consent. All data collected to be shared outside of the research team will be aggregated data for the purpose of publications.

REFERENCES:
- [Background] Bousquet B, Green MA, Caillouette CN, Simon J, Padwa BL, Resnick CM. How Much Opioid Medication Do Patients Need After Orthognathic Surgery? J Oral Maxillofac Surg. 2022 Jul;80(7):1174-1182. doi: 10.1016/j.joms.2022.04.002. Epub 2022 Apr 7. PMID 35526579
- [Background] Macintyre PE, Quinlan J, Levy N, Lobo DN. Current Issues in the Use of Opioids for the Management of Postoperative Pain: A Review. JAMA Surg. 2022 Feb 1;157(2):158-166. doi: 10.1001/jamasurg.2021.6210. PMID 34878527
- [Background] Pathan H, Williams J. Basic opioid pharmacology: an update. Br J Pain. 2012 Feb;6(1):11-6. doi: 10.1177/2049463712438493. PMID 26516461
- [Background] Borgland SL. Acute opioid receptor desensitization and tolerance: is there a link? Clin Exp Pharmacol Physiol. 2001 Mar;28(3):147-54. doi: 10.1046/j.1440-1681.2001.03418.x. PMID 11207668
- [Background] Kaye AD, Jones MR, Kaye AM, Ripoll JG, Galan V, Beakley BD, Calixto F, Bolden JL, Urman RD, Manchikanti L. Prescription Opioid Abuse in Chronic Pain: An Updated Review of Opioid Abuse Predictors and Strategies to Curb Opioid Abuse: Part 1. Pain Physician. 2017 Feb;20(2S):S93-S109. PMID 28226333
- [Background] Belzak L, Halverson J. The opioid crisis in Canada: a national perspective. Health Promot Chronic Dis Prev Can. 2018 Jun;38(6):224-233. doi: 10.24095/hpcdp.38.6.02. PMID 29911818
- [Background] Miech R, Johnston L, O'Malley PM, Keyes KM, Heard K. Prescription Opioids in Adolescence and Future Opioid Misuse. Pediatrics. 2015 Nov;136(5):e1169-77. doi: 10.1542/peds.2015-1364. PMID 26504126
- [Background] Lawal OD, Gold J, Murthy A, Ruchi R, Bavry E, Hume AL, Lewkowitz AK, Brothers T, Wen X. Rate and Risk Factors Associated With Prolonged Opioid Use After Surgery: A Systematic Review and Meta-analysis. JAMA Netw Open. 2020 Jun 1;3(6):e207367. doi: 10.1001/jamanetworkopen.2020.7367. PMID 32584407
- [Background] Clarke H, Soneji N, Ko DT, Yun L, Wijeysundera DN. Rates and risk factors for prolonged opioid use after major surgery: population based cohort study. BMJ. 2014 Feb 11;348:g1251. doi: 10.1136/bmj.g1251. PMID 24519537
- [Background] Tamboli M, Mariano ER, Gustafson KE, Briones BL, Hunter OO, Wang RR, Harrison TK, Kou A, Mudumbai SC, Kim TE, Indelli PF, Giori NJ. A Multidisciplinary Patient-Specific Opioid Prescribing and Tapering Protocol Is Associated with a Decrease in Total Opioid Dose Prescribed for Six Weeks After Total Hip Arthroplasty. Pain Med. 2020 Nov 7;21(7):1474-1481. doi: 10.1093/pm/pnz260. PMID 31710680
- [Background] Joo SS, Hunter OO, Tamboli M, Leng JC, Harrison TK, Kassab K, Keeton JD, Skirboll S, Tharin S, Saleh E, Mudumbai SC, Wang RR, Kou A, Mariano ER. Implementation of a patient-specific tapering protocol at discharge decreases total opioid dose prescribed for 6 weeks after elective primary spine surgery. Reg Anesth Pain Med. 2020 Jun;45(6):474-478. doi: 10.1136/rapm-2020-101324. Epub 2020 Mar 31. PMID 32238478
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Kukushliev VV, Sherman KA, Kurylo CM, Ortmann SD, Scheidt RA, Scheidt KB. Tapered Dose Postoperative Opioid Prescriptions Following Inpatient Total Hip and Knee Arthroplasty: Quality Improvement Study and Retrospective Review. J Arthroplasty. 2023 Feb;38(2):239-244. doi: 10.1016/j.arth.2022.08.043. Epub 2022 Sep 6. PMID 36075313
- [Background] Yajnik M, Hill JN, Hunter OO, Howard SK, Kim TE, Harrison TK, Mariano ER. Patient education and engagement in postoperative pain management decreases opioid use following knee replacement surgery. Patient Educ Couns. 2019 Feb;102(2):383-387. doi: 10.1016/j.pec.2018.09.001. Epub 2018 Sep 5. PMID 30219634
- [Background] Von Korff M, Saunders K, Thomas Ray G, Boudreau D, Campbell C, Merrill J, Sullivan MD, Rutter CM, Silverberg MJ, Banta-Green C, Weisner C. De facto long-term opioid therapy for noncancer pain. Clin J Pain. 2008 Jul-Aug;24(6):521-7. doi: 10.1097/AJP.0b013e318169d03b. PMID 18574361
- [Background] Precious DS, Multari J, Finley GA, McGrath P. A comparison of patient-controlled and fixed schedule analgesia after orthognathic surgery. J Oral Maxillofac Surg. 1997 Jan;55(1):33-9; discussion 40. doi: 10.1016/s0278-2391(97)90442-0. PMID 8994466
- [Background] Moerman N, van Dam FS, Muller MJ, Oosting H. The Amsterdam Preoperative Anxiety and Information Scale (APAIS). Anesth Analg. 1996 Mar;82(3):445-51. doi: 10.1097/00000539-199603000-00002. PMID 8623940
- [Background] Polomano RC, Galloway KT, Kent ML, Brandon-Edwards H, Kwon KN, Morales C, Buckenmaier C' 3rd. Psychometric Testing of the Defense and Veterans Pain Rating Scale (DVPRS): A New Pain Scale for Military Population. Pain Med. 2016 Aug;17(8):1505-19. doi: 10.1093/pm/pnw105. Epub 2016 Jun 6. PMID 27272528
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660